CLINICAL TRIAL: NCT02544607
Title: Baseline Insular Dysfunction as a Predictor of Ketamine's Antidepressant Effects in Anxious Depression
Brief Title: Ketamine for Depression: An MRI Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brain & Behavior Research Foundation (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Cristina Cusin, M.D., Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015P001912; 24032 (Other Grant/Funding Number: 2015 NARSAD Young Investigator Grant)
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Depression; Anxious Depression; Major Depressive Disorder
Keywords: Ketamine; Depression; Anxious Depression; MRI
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Ketamine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine + MRI (Experimental): All eligible participants will receive open label ketamine and undergo Magnetic Resonance Imaging (MRI).
  Interventions: Drug: Ketamine; Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: Ketamine — Ketamine 0.5mg/kg over 40 minutes IV
  Other Names: Ketamine Hydrochloride
Other: Magnetic Resonance Imaging (MRI) — MRI technology will be used before and after ketamine for patients with depression

SUMMARY:
Ketamine has been shown to decrease symptoms of anxious depression quickly. This decrease has been shown to last for up to one month. MRI technology will be used before and after ketamine for patients with depression to examine the extent to which certain brain areas predict ketamine's antidepressant effects.

DETAILED DESCRIPTION:
Ketamine's antidepressant effects were measured with Hamilton Depression Rating Scale (HDRS). MRI data will also be analyzed to examine the extent to which certain brain areas predict ketamine's antidepressant effects.

ELIGIBILITY:
Inclusion Criteria: Patients with Depression

Patients will:

1. be 18-64 years old,
2. read, understand, and provide written informed consent in English,
3. meet criteria for a primary psychiatric diagnosis of major depressive disorder for ≥ 4 weeks,
4. have a history of ≥1 failed medication trial during the current depression
5. be on a stable antidepressant and psychotherapy regimen for ≥28 days,
6. maintain a treating doctor who is in agreement with study participation,
7. have a reliable chaperone accompany them home following the completion of the ketamine infusion day,
8. be generally healthy, as assessed by medical history, physical examination (including vital signs), clinical laboratory evaluations, and electrocardiogram (EKG),
9. be of non-childbearing potential or use of an acceptable form of birth control (females only),
10. be right handed.

Exclusion Criteria: Patients with Depression

Patients will be excluded if any of the following criteria are met:

1) delirium or dementia diagnosis, 2) unstable medical illness or clinically significant laboratory results, 3) history of clinically significant cardiovascular disease or electrocardiogram (EKG) findings, or medical conditions that put the patient at risk for possible cardiac side effects or alter brain morphology (e.g., traumatic brain injury), 4) history of multiple adverse drug reactions, 5) current/past history of psychotic disorders, 6) active substance use disorders (except nicotine and caffeine) within the past six months or past history of ketamine/PCP abuse, 7) requirement of excluded medications that may interact with ketamine, 8) weigh >250 lbs., 9) pregnancy, breastfeeding, or unacceptable means of birth control (females only) 10) presence of MRI contraindications (e.g., presence of metallic (ferromagnetic) implants (e.g., heart pacemaker, aneurysm clips)), 11) current serious suicidal or homicidal risk, or 12) concurrent participation in other research studies.

---------------------------------------------------------------------------------------

Inclusion Criteria: Healthy Controls

Healthy Controls will:

1. be 18-64 years old,
2. read, understand, and provide written informed consent in English,
3. have a reliable chaperone accompany them home following the completion of the ketamine infusion day,
4. be generally healthy, as assessed by medical history, physical examination (including vital signs), clinical laboratory evaluations, and electrocardiogram (EKG),
5. be of non-childbearing potential or use of an acceptable form of birth control (females only), and
6. be right handed.

Exclusion Criteria: Healthy Controls

Healthy controls will be excluded if any of the following criteria are met:

1. current or past psychiatric diagnosis (excluding phobias), including alcohol or substance abuse or dependence diagnosis (except for nicotine or caffeine),
2. presence of MRI contraindications (e.g., presence of metallic (ferromagnetic) implants (e.g., heart pacemaker, aneurysm clips)),
3. presence of medical illness likely to alter brain morphology and/or physiology (e.g., traumatic brain injury),
4. requirement of excluded medications that may interact with ketamine,
5. presence of psychiatric disorders in first-degree relatives,
6. pregnancy, breastfeeding, or unacceptable means of birth control (females only), or
7. weight >250 lbs.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Cusin, M.D., Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MGH Depression Clinical and Research Program — http://www.depressionmgh.org/our-studies

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As specified, the total number of participants enrolled are those who agreed to participate in the study following completion of the informed consent process (n=25). This number does not reflect the number of subjects who actually started treatment (n=16).
Groups:
- Ketamine + MRI: All eligible participants will receive open label ketamine and undergo Magnetic Resonance Imaging
  Ketamine: Ketamine 0.5mg/kg over 40 minutes IV
Period: Overall Study
Arm/Group | Ketamine + MRI
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ketamine: All eligible participants will receive open label ketamine
  Ketamine: Ketamine 0.5mg/kg over 40 minutes IV
Arm/Group | Ketamine
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale (HDRS) From Baseline/Minute 0 to 4 Hours Post-infusion.
Description: Hamilton Depression Rating Scale; possible scores range from 0 to 81 with higher scores indicating higher depression symptoms
  Change will be calculated by difference between HDRS from Minute 0 to Minute 240.
Time Frame: 4 hours
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 16
score on a scale | -9.625 [-25 to 6]
Statistical Analysis 1: Comparison: Ketamine; Test type: Other; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Percent Change in Tissue Fractional Anisotropy Quantification (Left Inferior Longitudinal Fasciculus)
Description: Free-water imaging, a two-compartment diffusion model, was employed to quantify tissue fractional anisotropy (FAt) pre- and post-infusion
Time Frame: 4 hours
Population: Reasons for missing data (N=3) included a scanner malfunction and participant requests to stop scanning prior to dMRI sequence acquisition.
Measure: Number; unit: percent change
Arm/Group | Ketamine + MRI
Number analyzed (Participants) | 13
percent change | .901
Statistical Analysis 1: Comparison: Ketamine + MRI; Test type: Other; p = 0.048, t-test, 2 sided

3. Secondary Outcome: Percent Change in Tissue Fractional Anisotropy Quantification (Right Inferior Longitudinal Fasciculus)
Description: as for outcome 2
Time Frame: 4 hours
Population: as for outcome 2
Measure: Number; unit: percent change
Arm/Group | Ketamine + MRI
Number analyzed (Participants) | 13
percent change | 1.247
Statistical Analysis 1: Comparison: Ketamine + MRI; Test type: Other; p = 0.003, t-test, 2 sided

4. Secondary Outcome: Percent Change in Tissue Fractional Anisotropy Quantification (Left Superior Longitudinal Fasciculus)
Description: as for outcome 2
Time Frame: 4 hours
Population: as for outcome 2
Measure: Number; unit: percent change
Arm/Group | Ketamine + MRI
Number analyzed (Participants) | 13
percent change | .696
Statistical Analysis 1: Comparison: Ketamine + MRI; Test type: Other; p = .0499, t-test, 2 sided

5. Secondary Outcome: Percent Change in Tissue Fractional Anisotropy Quantification (Right Uncinate Fasciculus)
Description: as for outcome 2
Time Frame: 4 hours
Population: as for outcome 2
Measure: Number; unit: percent change
Arm/Group | Ketamine + MRI
Number analyzed (Participants) | 13
percent change | 1.158
Statistical Analysis 1: Comparison: Ketamine + MRI; Test type: Other; p = 0.038, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the course of the study. The collection of this data took place at the initial screen, continuously throughout the duration of the administration visit (e.g. Visit 2), 24 hours post-administration, and up to 3 months following the administration visit.
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine (N=16)
bilateral nystagmus (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT02544607/Prot_SAP_000.pdf